CLINICAL TRIAL: NCT06163547
Title: Middle Meningeal Artery (MMA) Embolization for cSDH: Rationale and Design for the STOp Recurrence of MMA Bleeding (STORMM) Randomized-Control Trial
Brief Title: Middle Meningeal Artery Embolization for Chronic Subdural Hematomas (STORMM)
Acronym: STORMM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Aria Nouri, Dr., University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-00848
Record Dates: First submitted 2023-11-20; First posted 2023-12-11 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Chronic Subdural Hematomas; Cerebral Compression Due to Injury
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Intervention Model Description: This study is a multicentre randomised-controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 - Surgery - No embolization (control) (No Intervention): Patients who undergo surgical treatment will be randomized into receiving embolization within 72 hours post-surgery (Arm 2) or no-embolization post-surgery (conventional management, Arm 1). Patients will be randomized at rate of 2 MMA embolization to 1 conventional management.
- Arm 2 - Surgery - MMA embolisation (Experimental): Patients who undergo surgical treatment will be randomized into receiving embolization within 72 hours post-surgery (Arm 2) or no-embolization post-surgery (conventional management, Arm 1). Patients will be randomized at rate of 2 MMA embolization to 1 conventional management.
  Interventions: Radiation: MMA embolization
- Arm 3 - No surgery - Embolization accepted (Active Comparator): Patients who are excluded for surgery due to significant medical contraindications or patients who refuse surgery, will be considered for embolization only. Embolization accepted : Arm 3.
  Interventions: Radiation: MMA embolization
- Arm 4 - No surgery - Embolization not accepted (No Intervention): Patients who are excluded for surgery due to significant medical contraindications or patients who refuse surgery, will be considered for embolization only. Embolization refused : Arm 4.

INTERVENTIONS:
Radiation: MMA embolization — Middle meningeal artery embolization
  Arms: Arm 2 - Surgery - MMA embolisation; Arm 3 - No surgery - Embolization accepted

SUMMARY:
Chronic Subdural Hematomas (cSHD) are common, and due to cerebral compression, often result in neurological impairment and reduced consciousness. Surgery is typically performed once neurological symptoms develop. Recent studies suggest that arteries nourished by the middle meningeal artery (MMA) may be responsible for hematoma progression and that MMA embolization is clinically useful. There is less evidence, that embolization of MMA also may be a treatment option for individuals without surgical treatment. The investigators propose a multicentre study to investigate both potentials: (1) Assessment of efficacy of embolization after surgery to reduce recurrence and improve outcomes by conducting a randomized trial (randomization arms; Arms 1 and 2), (2) Assessment of embolization-alone efficacy when surgery is contraindicated or refused (embolization-only arm, Arms 3 and 4).

DETAILED DESCRIPTION:
Evidence to support the benefit of MMA embolization remains limited and the risk-benefit balance remains unclear. Case series have shown that recurrence rates with embolization are much lower, and that embolization is generally very safe. Risks associated with neurointerventional procedures will be directly discussed with patients or their caretakers as part of the conventional consenting procedure. Risks include access site hematoma, radiation exposure, vascular injury, brain ischemia, death (theoretic and extremely unlikely) and typical risks associated with general or local anaesthesia. The potential efficacy of MMA embolization as a treatment therefore requires higher level evidence in the form of randomized control trials.

The benefit of the embolization is a substantial reduction in recurrence of cSDH, which has been reported to be as high 1 in 3-4 patients. Recurrence of cSDH can lead to additional surgery and complications.

First objective: Evaluate the recurrence rates of cSDH after combined surgical and MMA embolization treatments (Arm 2) versus surgery alone (Arms 1).

Second objective: The second objective is to evaluate the stability and regression of cSDH after for all the Arms of the study at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-100
* Consent possible
* cSDH located at the convexities
* Patients with symptomatic cSDH
* Patients with asymptomatic large chronic/subacute hematoma after 6 weeks of failed conservative treatment

Exclusion Criteria:

* Consent not possible
* Pregnancy
* Prisoner
* Angiography contraindication
* Patient for whom follow-up is problematic (e.g. distant residency, homeless …)
* Previous surgery for cSDH

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence of cSDH - 1 | 6-months
  Surgical reoperation
Recurrence of cSDH - 2 | 6-months
  Neurological deterioration due to a cSDH after evacuation
Recurrence of cSDH - 3 | 6-months
  Post-operative hematoma volume of more than 90% of the preoperative volume at follow-up

SECONDARY OUTCOMES:
Additional clinical outcomes - 1 | 6-months
  Glasgow Coma Scale (Min=3; Max=15; Higher score=Best outcome)
Additional clinical outcomes - 2 | 6-months
  modified Ranking Scale (Min=0; Max=6; Higher score=Worse outcome)
Additional clinical outcomes - 3 | 6-months
  Markwalder Grading Scale (Min=0; Max=4; Higher score=Worse outcome)
Additional clinical outcomes - 4 | 6-months
  Glasgow Outcome Scale - Extended (Min=1; Max=8; Higher score=Best outcome)
Additional clinical outcomes - 5 | 6-months
  Karnofsky Performance Score (Min=20; Max=100; Higher score=Best outcome)
Additional clinical outcomes - 6 | 6-months
  Therapy-Disability-Neurology grading system (Min=1; Max=5; Higher score=Worse outcome)
Additional clinical outcomes - 7 | 6-months
  Mortality rate
Additional clinical outcomes - 8 | 6-months
  Re-hospitalisation for all causes

CONTACTS AND LOCATIONS:
Overall Officials: Aria Nouri, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al Awadhi A, Mollica C, Da Broi M, Molliqaj G, Hofmeister J, Rosi A, Bernava G, Machi P, Morel S, Cardia A, Meling TR, Schaller K, Nouri A. Middle meningeal artery (MMA) embolisation for chronic subdural haematomas: rationale and design for the STOp Recurrence of MMA Bleeding (STORMM) randomised control trial-a study protocol. BMJ Open. 2025 May 6;15(5):e092014. doi: 10.1136/bmjopen-2024-092014. PMID 40335147

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT06163547/Prot_SAP_002.pdf